CLINICAL TRIAL: NCT04145505
Title: Influence of the Presence of Ganglionar Micrometastases Associated With an Elevation of Angiogenesis on the Evolution of Colon Cancer. Prognostic Value of the Levels of VEGF-A Anf VEGF-C
Brief Title: Micrometastases and Angiogenesis in Colon Cancer. Prognostic Value of VEGF.
Acronym: VEGF-GC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, M. Carmen Balague Ponz, Principal investigator, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Other Study IDs: IIBSP-VEG-2018-77
Record Dates: First submitted 2019-10-26; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Colorectal Cancer; Angiogenesis
Keywords: SENTINEL NODE
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood + tumor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: COLORECTAL CANCER SURGERY — SENTINEL NODE DETECTION

SUMMARY:
According to current clinical guidelines adjuvant treatment in colon cancer is not recommended in patients with stage I and IIA, and in patients with high risk factors (IIB) adjuvant treatment has not shown a clear benefit in recurrence or survival.

However, more than 20% of these patients have recurrence. This high percentage raises the possible understaging of current methods, so in recent years different methods have been developed in order to obtain a correct staging that have allowed a greater detection of micrometastasis (less than 2mm).

The performance of the detection technique of the sentinel node in colon cancer allows us to perform this study in 1-3 lymph nodes, so that performing in all the nodes removed in a piece would be imposible in daily clinical practice for time, personnel and economic resources needed to do it.

This technique achieves between 5-15% of overstaging which means that in stages I and IIA can lead to a change in the indication of adjuvant treatment. Despite this, the influence of ganglion micrometastases on survival is still controversial. This leads to consider other factors that may influence tumor aggressiveness, such as an increase in angiogenesis that allows the viability of implants less than 2mm. Therefore, we propose that elevated levels of VEGF (angiogenesis marker) in patients with sentinel lymph node micrometastases can lead to a worse prognosis.

Based on these premises, the aim of the study is to assess the correlation between the levels of serum and tumor VEGF-A and VEGF-C (markers of angiogenesis and lymphangiogenesis) and the evolution of the disease in patients with lymph node micrometastases.

DETAILED DESCRIPTION:
Once the investigators have all the data of the patients included in the study, and the ELISA analysis of the serum and tissue VEGF levels has been performed, we hope to determine a threshold level of VEGF in blood and tissue that modifies the prognostic implications of the presence of ganglionic micrometastasis, which increases the viability of these implants.

If the investigators determine this threshold and demonstrate that high levels of this molecule, both in blood and tissue, increase the rate of recurrence in patients with lymph node micrometastases, would be suggested a change in the indications for adjuvant treatment in patients in whom it is not currently indicated (stages I-IIA and IIB without other factors of poor prognosis) considering that they have an independent bad prognostic factor such as a high level (above our threshold) of VEGF. This allows the investigators to select those patients who would benefit from chemotherapy treatment despite not being indicated according to the current treatment guidelines (NCCN 2018).

ELIGIBILITY:
Inclusion criteria:

* Patients older than 18 years
* Diagnosis of colon adenocarcinoma located above promontory
* Elective surgical treatment with oncological criteria and curative intention

Exclusion criteria:

* Non-acceptance by the patient
* Patients who have received QT during the preoperative period
* Patients with previous colon surgery
* Patients with definitive study of the surgical piece with involvement of the lymph nodes according to conventional histological study (Stage III)
* Patients presenting distant dissemination in the extension study (Stage IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with colonic cancer and curative surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-26 (Actual); Primary Completion 2020-02-21 (Estimated); Study Completion 2021-02-21 (Estimated)

PRIMARY OUTCOMES:
recurrence | 5 years
  local, lymph node or distant mtastasis appearance

CONTACTS AND LOCATIONS:
Overall Officials: CARMEN BALAGUÉ PONS, PHD DR, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No